CLINICAL TRIAL: NCT03848247
Title: The Effect of Experimental Neck Pain in Healthy Participants - The Transition From Acute to Ongoing Pain
Brief Title: The Effect of Experimental Neck Pain in Healthy Participants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Steffan Wittrup Christensen, Assistant professor, Aalborg University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: N-20180063_Sub-project_1
Record Dates: First submitted 2019-02-16; First posted 2019-02-20 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Healthy; Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Experimental): Participants will be injected with 0.5ml Isotonic saline into a neck muscle
  Interventions: Other: Injection of Isotonic saline
- Neck pain (Experimental): Participants will be injected with 0.5ml NGF into the a neck muscle
  Interventions: Other: Injection of NGF

INTERVENTIONS:
Other: Injection of Isotonic saline — Half the participants will be injected in a neck muscle with isotonic saline (Control group) and the other half will get NGF (Neck pain group).
  Arms: Control group
Other: Injection of NGF — Half the participants will be injected in a neck muscle with NGF (Neck pain group).
  Arms: Neck pain

SUMMARY:
This study investigates if/how an experimentally applied muscle pain/soreness, lasting for some days may affect brain activity, balance, movement patterns, muscle function and pain sensitivity in a healthy population

DETAILED DESCRIPTION:
All included healthy volunteers will participate in test-sessions on 4 separate days over approximately 2 weeks.

During the study participants will be randomised into and either a control group (injection of isotonic saline into a neck muscle) or neck pain group (injection of Nerve Growth Factor (NGF) into a neck muscle).

Alle participants tested with regards to:

Brain activity related to neck muscles will be estimated using TMS Balance will be tested using a force place Body movements will be recorded using 3D tracking Muscle activity will be estimated using electromyography (EMG)

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women aged 18-50 years
* Only for sub-projects 1 and 2: Right-handed
* Able to speak, read and understand Danish and English

Exclusion Criteria:

* Pain from the neck or shoulder area during the past 6 months
* Experience of delayed onset muscle soreness (DOMS) during the week leading up to the test session
* Former surgery in neck or shoulder
* Current or previous chronic or recurrent pain condition
* Pregnancy
* Drug addiction defined as the use of cannabis, opioids or other drugs
* Previous neurologic, musculoskeletal or mental illnesses
* Regular use of analgesics
* Abnormally disrupted sleep in the last 24 hours preceding the experiment
* Lack of ability to cooperate
* Unable to pass the TASS safety screening questionnaire for TMS

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-01-21 (Actual); Primary Completion 2019-05-01 (Estimated); Study Completion 2019-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in pressure pain threshold (PPT) measured with a handheld pressure algometer | Day 0, 2,4 and 15
  PPT will be assessed over head, neck, arm and leg sites.
Change in motor evoked potentials | Day 0, 4 and 15
  Trans cranial magnetic stimulation (TMS) is used to asses motor evoked potentials of neck muscles
Change in Body movement | Day 0, 4 and 15
  3D recordings of body movements

SECONDARY OUTCOMES:
Change in muscle activity (EMG) | Day 0, 4 and 15
  EMG of axioscapular muscles & trunk during arm movements
Change in standing balance | Day 0, 4 and 15
  Standing balance is measured on a force platform
Change in perceived pain: McGill Pain Questionnaire | Day 0, 2,4 and 15
  Pain will be scored using a scale from 0-10 with 0 being no pain and 10 being worst imaginable pain, by drawing on body charts and choosing words from the McGill Pain Questionnaire.
Disability | Day 0, 2,4 and 15
  Neck disability Index will be scored. Body movements will be scored on a modified 6-point Likert scale (0 = not difficult at all; 1 = minimally difficult; 2 = somewhat difficult; 3 = fairly difficult; 4 = very difficult; 5 = unable to perform)
Pain Catastrophizing Scale (13 item questionnaire) | Day 2
  Pain Catastrophizing Scale (PCS) questionnaire. 13 items that can be answered with a Likert scale (0 = not at all, 1 = to a slight degree, 2= to a moderate degree, 3 = to a great degree, 4 = all the time).
  The PCS is scored by summing responses to all 13 items with scores ranging from 0 - 52.
The Big Five Inventory (BFI) | Day 2
  BFI questionnaire investigates five general traits personality: extraversion, agreeableness, conscientiousness, neuroticism and openness. The BFI consists of 44 items that are answered on a 5 point Likert scale (1=Disagree strongly, 2=Disagree a little, 3=Neither agree or disagree, 4=Agree a little, 5=Agree strongly). This is not good/bad score in this questionnaire as it only assess personality traits.

CONTACTS AND LOCATIONS:
Overall Officials: Steffan W Christensen, PhD, Principal Investigator — Aalborg University
Locations (1):
- Dept. Of Health Science and Technology, SMI, Aalborg University, Aalborg, Denmark

REFERENCES:
- [Derived] Simonsen MB, Cancino EE, de Brito Silva P, Sorensen LB, Hirata RP, Christensen SWM. The impact of prolonged experimental neck pain on walking stability and gait kinematics - A parallel-group study. Clin Biomech (Bristol). 2023 Jan;101:105869. doi: 10.1016/j.clinbiomech.2022.105869. Epub 2022 Dec 23. PMID 36584579